CLINICAL TRIAL: NCT01897649
Title: Effect of 15g Daily Consumption of NUTRIOSE During 2 and 4 Weeks on Healthy Volunteers Microbiota and Digestive Tolerance.
Brief Title: Effect of 15g Daily Consumption of NUTRIOSE on Healthy Volunteers Microbiota.
Acronym: ROQ_NUTRIFLORE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nealth Sarl (Network)
Collaborators: Roquette Freres (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ROQ_NUTRIFLORE10
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Microbiota; Dietary Fibers
Keywords: functional food; digestive tolerance; microbiota; bifidogenic effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NUTRIOSE (Experimental): group of volunteers fed with NUTRIOSE
  Interventions: Dietary Supplement: NUTRIOSE FB06
- GLUCIDEX (Active Comparator): gruop of volunteers fed with GLUCIDEX
  Interventions: Dietary Supplement: GLUCIDEX 21

INTERVENTIONS:
Dietary Supplement: NUTRIOSE FB06 — 15g/day NUTRIOSE FB06
  Arms: NUTRIOSE
Dietary Supplement: GLUCIDEX 21 — 15g/day GLUCIDEX 21
  Arms: GLUCIDEX

SUMMARY:
NUTRIOSE is a food ingredient defined as a carbohydrate polymer of vegetable origin (wheat starch or corn) with a degree of polymerization ≥ 3 and chemically transformed. It is soluble in aqueous solution, very poorly digested in the small intestine, it mostly reaches the colon where it stimulates fermentation. AFSSA, in its opinion of July 30, 2007, considers that this ingredient is a "soluble dietary fiber." The objective of this research is to determine, among healthy subjects, the effect of this dietary fiber on changes in gut microbiota and digestive tolerance during a 28 days consumption. Microbiological analyzes will be performed by RT-PCR. Digestive tolerance will be measured by the intelligence of a questionnaire by volunteers.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 50 years,
* BMI 18 to 25 kg/m2,
* absence of known or scalable organic or psychiatric disease
* no history of chronic gastrointestinal disease
* having a bowel regularity (1-3 defecation per day, of normal consistency),
* person without medication during the study (especially laxatives, anti diarrheal) (except contraceptives in women)
* having normal laboratory hepatic and renal tests (ASAT, ALAT, GGT, urea, creatinine)
* no pregnant nor nursing women
* covered by Social Security
* negative serology for hepatitis B/C and HIV
* who signed the informed consent form

Exclusion Criteria:

* persons abusing drugs (laxatives, anti-diarrheal)
* person who doesn't want to stop taking food supplements containing pre- or probiotics during time of the study
* person intolerant to gluten and / or allergic to wheat flour
* person in vegetarian or vegan diet
* Inclusion in another clinical study
* subjects receiving over 4,500 Euros in the last 12 months (including the present study)
* subjects presenting risk of non-compliance in the opinion of the recruiting doctor.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Clostridium Perfringens rate in stool | D0 ; D14 ; D28

SECONDARY OUTCOMES:
digestive tolerance | J0 to J28 (every day)
stool pH | D0 ; D14; D28
total stool flora | D0 ; D14 ; D28
Bacteroides rate in stool | D0 ; D14 ; D28
Eubacterium rectal rate in stool | D0 ; D14 ; D28
Clostridium coccoides rate in stool | D0 ; D14 ; D28
Clostridium leptum rate in stool | D0 ; D14 ; D28
Bifidobacteria rate in stool | D0 ; D14 ; D28
Lactobacteria rate in stool | D0 ; D14 ; D28
Streptococcus rate in stool | D0 ; D14 ; D28
Enterococcus rate in stool | D0 ; D14 ; D28
Bacteroidetes rate in stool | D0 ; D14 ; D28
Actinobacteria rate in stool | D0 ; D14; D28
Firmicutes rate in stool | D0 ; D14 ; D28
E. Coli rate in stool | D0 ; D14 ; D28
Clostridium difficile rate in stool | D0 ; D14 ; D28
Faecalibacterium prausnitzii rate in stool | D0 ; D14 ; D28
Clostridium difficile typa A and B rate in stool | D0 ; D14 ; D28
E. Coli EIEC + EPEC (eae gene) rate in stool | D0 ; D14 ; D28
Shigella + E. Coli EIEC (ipaH gene) rate in stool | D0 ; D14 ; D28
Listeria Monocytogenes rate in stool | D0 ; D14 ; D28
Yersinia Enterocolitica rate in stool | D0 ; D14 ; D28

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, MD,PhD, Principal Investigator — Centre de Recherche en Nutrition Humaine d'Ile-de-France
Locations (1):
- Hopital Avicenne- Centre de Recherche Sur Volontaires-Service de Gastroenterologie, Bobigny, France

REFERENCES:
- [Background] Li S, Guerin-Deremaux L, Pochat M, Wils D, Reifer C, Miller LE. NUTRIOSE dietary fiber supplementation improves insulin resistance and determinants of metabolic syndrome in overweight men: a double-blind, randomized, placebo-controlled study. Appl Physiol Nutr Metab. 2010 Dec;35(6):773-82. doi: 10.1139/H10-074. PMID 21164548
- [Background] Guerin-Deremaux L, Li S, Pochat M, Wils D, Mubasher M, Reifer C, Miller LE. Effects of NUTRIOSE(R) dietary fiber supplementation on body weight, body composition, energy intake, and hunger in overweight men. Int J Food Sci Nutr. 2011 Sep;62(6):628-35. doi: 10.3109/09637486.2011.569492. Epub 2011 May 19. PMID 21591985
- [Background] Pasman W, Wils D, Saniez MH, Kardinaal A. Long-term gastrointestinal tolerance of NUTRIOSE FB in healthy men. Eur J Clin Nutr. 2006 Aug;60(8):1024-34. doi: 10.1038/sj.ejcn.1602418. Epub 2006 Feb 15. PMID 16482066
- [Background] Haarman M, Knol J. Quantitative real-time PCR assays to identify and quantify fecal Bifidobacterium species in infants receiving a prebiotic infant formula. Appl Environ Microbiol. 2005 May;71(5):2318-24. doi: 10.1128/AEM.71.5.2318-2324.2005. PMID 15870317